CLINICAL TRIAL: NCT03336463
Title: Prediction of Recurrent Pregnancy Loss by a New Thrombophilia Based Genetic Risk Score
Acronym: TiC-RPL
Status: Completed | Type: Observational
Sponsor: Ferrer inCode, S.L. (Industry)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other); Instituto de Salud Carlos III (Other Government); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Instituto Valenciano de Infertilidad, IVI VALENCIA (Other); IVI-RMA London (Unknown); Instituto de Investigacion Sanitaria La Fe (Other); Gendiag.exe, S.L. (Unknown); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: FerrerinCode
Record Dates: First submitted 2017-10-23; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Miscarriage, Recurrent
Keywords: Thrombophilia screening; Genetic risk score
MeSH Terms: conditions — Abortion, Habitual; Genetic Risk Score

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA extraction from saliva or blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: No intervention
- Cases: No intervention

SUMMARY:
Recurrent pregnancy loss (RPL) is a clinical problem affecting 1-5% of couples of reproductive age. The contribution of thrombophilia to RPL is disputed. This controversy is partly due to low sensitivity of the genetic variants currently used to evaluate hereditary thrombophilia: the Leiden mutation (identified as rs6025) in the coagulation factor 5 (F5L) gene and mutation G20210A (identified as rs1799963) in the prothrombin (PT) gene.

Our objective was to determine whether a wider algorithm that includes clinic and genetic variants associated with thrombophilia could be more useful in the prediction for RPL than FVL and PT alone.

DETAILED DESCRIPTION:
Recurrent pregnancy loss can affect up to 5% of women in child-bearing age and is considered one of the most common causes of female sterility. In recent years, the association between thrombophilia and pregnancy failure has been observed in a number of studies, varying according to the nature of the thrombophilia (for example the antiphospholipid syndrome as opposed to the hereditary forms) or the type of pregnancy loss (either isolated or recurrent, or early or late). It has therefore been accepted that thrombophilia is detected in a significant number of idiopathic pregnancy losses, reaching 66% of the cases in some series.

Since the 1990's, a number of studies have associated recurrent pregnancy loss with FVL mutations (most frequently) and G20210 PT. In a systematic review, it was confirmed that women with thrombophilia have a higher risk of developing thromboembolism and complications in pregnancy. Another recent meta-analysis of prospective cohort studies concluded that women who were carriers of FVL had a higher risk of late pregnancy loss, at 52%, as opposed to non-carriers (OR=1.52), though the differences in absolute risk were discreet (4.2% and 3.2%, respectively). However, the analysis of these 2 single nucleotide polymorphisms (SNPs) showed low discriminative capacity and diagnostic sensitivity.

This study hypothesize that the use of the Thrombo inCode® in the screening for hereditary thrombophilia in patients with recurrent pregnancy loss can improve the diagnostic sensitivity and predictive capacity of the routine genetic panel, based on FVL and G20210A PT. Thus, the Thrombo inCode® model can accurately identify more patients with clinical-genetic risk of thromboembolism and therefore establish the appropriate preventive measures.

A transversal observational case-control study will be carried out, with retrospective data analysis. The screening for hereditary thrombophilia will be performed through the Thrombo inCode® panel in cases and controls. The results produced from a single genetic analysis will allow comparison to the centres' routine protocol (FV Leiden and G20210A PT) with the complete Thrombo inCode® panel, that also includes the previously-mentioned classical variants.

ELIGIBILITY:
CONTROLS

Inclusion Criteria:

* Women >18 and < 38 years old at the time of the first pregnancy.
* Women with successful implantation and at least one full-term pregnancy
* No chronic pathology

Exclusion Criteria:

* Personal or family history of thrombosis
* Personal history of obstetric complications Miscarriage or foetal death Pre-eclampsia or eclampsia Intrauterine growth restriction Placental abruption
* Concomitant anticoagulant treatment and/or antiplatelet treatments during pregnancy

CASES

Inclusion Criteria:

* Repeated clinical miscarriages and/or foetal death (≥ 2 consecutive or ≥ 3 non- consecutive) before the 20th weeks of pregnancy, from spontaneous or assisted pregnancies.
* Recurrent miscarriage with the same gametic origin.

Idiopathic origin:

Women < 38 years old Non-severe seminal factor (sperm concentration > 2 mill/ml) Normal karyotypes in both spouses (or in the male and the donor in the case of ovocyte donation) Antiphospholipid syndrome negative Normal or corrected thyroid function BMI < 30

Exclusion Criteria:

* Diabetes
* Chronic pathologies
* Hydrosalpinx
* Concomitant anticoagulant or antiplatelet treatment

Ages: 18 Years to 37 Years | Sex: Female
Age Groups: Adult
Study Population: The study will include women with recurrent pregnancy loss (> 2 consecutive or > 3 non-consecutive) before the 20th week of pregnancy (cases) and women with at least 1 pregnancy at term (controls).
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Recurrent Pregnancy Loss | 20 weeks
  Repeated clinical pregnancy loss and/or foetal death (≥ 2 consecutive or ≥ 3 non-consecutive) before the 20th weeks of pregnancy
Pregnancy at term | 20 weeks
  Pregnancy with life-birth

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo S Salas, MD, PhD, Study Director — Ferrer inCode, S.L.
Locations (8):
- Spain (7):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Gendiag.exe, S.L., Esplugues de Llobregat, Select State
  - Institut d'Investigació Sant Pau, Barcelona
  - Instituto Salud Carlos III, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - IVI-RMA Valencia, Valencia
  - Instituto de Investigaciones Sanitarias La Fe, Valencia
- IVI-RMA-London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Soria JM, Morange PE, Vila J, Souto JC, Moyano M, Tregouet DA, Mateo J, Saut N, Salas E, Elosua R. Multilocus genetic risk scores for venous thromboembolism risk assessment. J Am Heart Assoc. 2014 Oct 23;3(5):e001060. doi: 10.1161/JAHA.114.001060. PMID 25341889